CLINICAL TRIAL: NCT03444818
Title: A Phase I, Open-label, Study to Determine the Absorption, Metabolism, and Excretion of [14C]-E6007 After a Single Oral Administration in Healthy Male Subjects
Brief Title: A Study to Determine the Absorption, Metabolism, and Excretion of [14C]-E6007 After a Single Oral Administration in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E6007-CP3; 2017-004119-38 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-02

CONDITIONS: Healthy Male Participants
Keywords: E6007; Pharmacokinetics; Radioactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-E6007 (Experimental): Participants will receive a single oral dose of 60 milligrams (mg) of [14C]-E6007.
  Interventions: Drug: [14C]-E6007

INTERVENTIONS:
Drug: [14C]-E6007 — Oral administration

SUMMARY:
This study will be conducted to evaluate the absorption, metabolism, and excretion of a single oral dose of [14C]-E6007 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 55 years of age
* Body mass index between 18.5 and 30.0 kilograms per meters squared (kg/m^2), and a total body weight between 50 and 100 kilograms (kg)
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead electrocardiogram, vital sign measurements, and clinical laboratory evaluations
* Males will agree to use contraception
* Able to comprehend and willing to sign an informed consent form and to abide by the study restrictions

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, and hernia repair will be allowed)
* Significant history or clinical manifestation of hemorrhoids
* History of alcoholism or drug/chemical abuse within 2 years prior to Check-in
* Positive hepatitis panel and/or positive human immunodeficiency virus test
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to Check-in
* Use or intend to use any prescription medications/products within 14 days prior to Check-in
* Participants in receipt of a live vaccine within 30 days prior to the first dose administration or who plan to receive a live vaccine during the study and for 14 days after the dose of study drug
* Use of tobacco or nicotine containing products within 3 months prior to Check-in
* Receipt of blood products within 2 months prior to Check-in
* Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening
* Participants with exposure to significant diagnostic or therapeutic radiation or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in
* Participants who have participated in any clinical trial involving a radiolabelled investigational product within 12 months prior to Check-in

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of E6007 derived from whole blood | Predose and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose
Area under the concentration-time curve (AUC) from time zero to infinity (AUC[0-∞]) postdose of E6007 | Predose and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose
Total radioactivity derived from whole blood | Up to 11 days
Total radioactivity in urine | Up to 11 days
Total radioactivity in feces | Up to 11 days

SECONDARY OUTCOMES:
Number of participants with any serious adverse event | Up to 11 days
Number of participants with any non-serious adverse event | Up to 11 days

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, West Yorkshire, United Kingdom